CLINICAL TRIAL: NCT02254824
Title: Effects and Underlying Mechanism of Lipid Lowering Intervention on Vascular Protection in Hypertensive Patients (EMINENT Study)
Brief Title: Effects and Underlying Mechanism of Lipid Lowering Intervention on Vascular Protection in Hypertensive Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: Peking University First Hospital (Other); Peking Union Medical College Hospital (Other); Beijing Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Aimin Dang, Cardiovascular Institute & Fuwai Hospital, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SF2011-4003-04
Record Dates: First submitted 2014-04-17; First posted 2014-10-02 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
Keywords: Xuezhikang; atorvastatin
MeSH Terms: conditions — Hypertension | interventions — xuezhikang; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Normal-dose statin (Active Comparator): Lifestyle modification with Normal-dose statin
  Interventions: Drug: Atorvastatin; Behavioral: Lifestyle modification
- Lifestyle modification + Xuezhikang (Active Comparator): Lifestyle changes with Xuezhikang
  Interventions: Drug: Xuezhikang; Behavioral: Lifestyle modification
- Lifestyle modification (Active Comparator): Lifestyle modification
  Interventions: Behavioral: Lifestyle modification

INTERVENTIONS:
Drug: Xuezhikang — Xuezhikang
  Arms: Lifestyle modification + Xuezhikang
Drug: Atorvastatin — Atorvastatin
  Arms: Normal-dose statin
Behavioral: Lifestyle modification — Lifestyle modification

SUMMARY:
The purpose of EMINENT study is to evaluate the efficacy of Xuezhikang or atorvastatin in hypertensive patients at low/moderate cardiovascular risk.

DETAILED DESCRIPTION:
EMINENT study is to evaluate the efficacy of Xuezhikang or atorvastatin on vascular function protection in hypertensive patients at low/moderate cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* All patients must meet the hypertension with low or moderate cardiovascular risk following 2010 Guidelines for prevention and treatment of hypertension in China

Exclusion Criteria:

* Secondary Hypertension
* Women who are pregnant or lactating
* History of mental instability, or major psychiatric illness not adequately controlled and stable on therapy
* Type 2 Diabetes
* Active liver disease or impaired liver function tests
* Impaired renal function
* Uncontrolled cardiac arrhythmia
* Patient who is unable to give informed consent
* Any condition or situation, which in the opinion of the investigator, might pose a risk to the patient or confound the results of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the Flow Mediated Dilatation (FMD) | 1 year

SECONDARY OUTCOMES:
the carotid - femoral Pulse Wave Velocity (cf-PWV), | 1 year
inflammatory markers | 1 year
lipid profiles | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Aimin Dang, Doctor, Principal Investigator — Fuwai Hospital & Cardiovascular Institute
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China